CLINICAL TRIAL: NCT07065578
Title: Optimization of the STAR Intervention on Self-care Symptom Management in Patients With Heart Failure
Brief Title: Optimization of STAR
Acronym: STAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Principal Investigator, H.Westland, Dr., UMC Utrecht
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 25u-0131; 03-004-2023-01 (Other: Dutch Heart Foundation)
Record Dates: First submitted 2025-06-19; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III
Keywords: Heart Failure; Self-management; symptom management; Self-care; e-Health
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This study has a randomized factorial experimental design with 2^3 = 8 experimental conditions to examine the effects of the three individual key modules. With this design, the main effects of each module and the interaction between modules will be tested. After informed consent, participants will be randomized using stratified block randomization to one of the eight experimental conditions within each participating HF clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Condition 1 (Experimental): Module 1: Low version; Module 2: Low version; Module 3: Low version
  Interventions: Other: STAR condition 1
- Condition 2 (Experimental): Module 1: Low version; Module 2: Low version; Module 3: High version
  Interventions: Other: STAR condition 2
- Condition 3 (Experimental): Module 1: Low version; Module 2: High version; Module 3: High version
  Interventions: Other: STAR condition 3
- Condition 4 (Experimental): Module 1: Low version; Module 2: High version; Module 3: Low version
  Interventions: Other: STAR condition 4
- Condition 5 (Experimental): Module 1: High version; Module 2: Low version; Module 3: Low version
  Interventions: Other: STAR condition 5
- Condition 6 (Experimental): Module 1: High version; Module 2: Low version; Module 3: High version
  Interventions: Other: STAR condition 6
- Condition 7 (Experimental): Module 1: High version; Module 2: High version; Module 3: Low version
  Interventions: Other: STAR condition 7
- Condition 8 (Experimental): Module 1: High version; Module 2: High version; Module 3: High version
  Interventions: Other: STAR condition 8

INTERVENTIONS:
Other: STAR condition 1 — * Basic module: HF information and doing symptom awareness exercises.
  * Low version Module 1: Symptom awareness exercises 2 times in 1 week, and written feedback HF nurse
  * Low version Module 2: Coaching in symptom management response and choose symptom response option to experiment with. Written feedback from HF nurse
  * Low version Module 3: Instruction and doing symptom management experiments for 2 weeks + keep logs; Written feedback HF nurse
  Arms: Condition 1
Other: STAR condition 2 — Basic module: aims to improve the participant's illness perceptions and standardize HF knowledge at the start of the intervention and doing exercises.- Low version Module 1: Symptom awareness exercises 2 times in 1 week, and written feedback HF nurse - Low version Module 2: Coaching in symptom management response and choose symptom response option to experiment with. Written feedback from HF nurse - High version Module 3: Instruction and doing symptom management experiments for 2 weeks + keep logs; Verbal feedback HF nurse
  Arms: Condition 2
Other: STAR condition 3 — Basic module: aims to improve the participant's illness perceptions and standardize HF knowledge at the start of the intervention and doing exercises.- Low version Module 1: Symptom awareness exercises 2 times in 1 week, and written feedback HF nurse - High version Module 2: Coaching in symptom management response and choose symptom response option to experiment with. Verbal feedback from HF nurse - High version Module 3: Instruction and doing symptom management experiments for 2 weeks + keep logs; Verbal feedback HF nurse
  Arms: Condition 3
Other: STAR condition 4 — Basic module: aims to improve the participant's illness perceptions and standardize HF knowledge at the start of the intervention and doing exercises.- Low version Module 1: Symptom awareness exercises 2 times in 1 week, and written feedback HF nurse - High version Module 2: Coaching in symptom management response and choose symptom response option to experiment with. Verbal feedback from HF nurse - Low version Module 3: Instruction and doing symptom management experiments for 2 weeks + keep logs; Written feedback HF nurse
  Arms: Condition 4
Other: STAR condition 5 — Basic module: aims to improve the participant's illness perceptions and standardize HF knowledge at the start of the intervention and doing exercises.- High version Module 1: Symptom awareness exercises 6 times in 2 weeks, and verbal feedback HF nurse - Low version Module 2: Coaching in symptom management response and choose symptom response option to experiment with. Written feedback from HF nurse - Low version Module 3: Instruction and doing symptom management experiments for 2 weeks + keep logs; written feedback HF nurse
  Arms: Condition 5
Other: STAR condition 6 — Basic module: aims to improve the participant's illness perceptions and standardize HF knowledge at the start of the intervention and doing exercises.- High version Module 1: Symptom awareness exercises 6 times in 2 weeks, and verbal feedback HF nurse - Low version Module 2: Coaching in symptom management response and choose symptom response option to experiment with. Written feedback from HF nurse - High version Module 3: Instruction and doing symptom management experiments for 2 weeks + keep logs; Verbal feedback HF nurse
  Arms: Condition 6
Other: STAR condition 7 — Basic module: aims to improve the participant's illness perceptions and standardize HF knowledge at the start of the intervention and doing exercises.- High version Module 1: Symptom awareness exercises 6 times in 2 weeks, and verbal feedback HF nurse - High version Module 2: Coaching in symptom management response and choose symptom response option to experiment with. Verbal feedback from HF nurse - Low version Module 3: Instruction and doing symptom management experiments for 2 weeks + keep logs; Written feedback HF nurse
  Arms: Condition 7
Other: STAR condition 8 — Basic module: aims to improve the participant's illness perceptions and standardize HF knowledge at the start of the intervention and doing exercises.- High version Module 1: Symptom awareness exercises 6 times in 2 weeks, and verbal feedback HF nurse - High version Module 2: Coaching in symptom management response and choose symptom response option to experiment with. Verbal feedback from HF nurse - High version Module 3: Instruction and doing symptom management experiments for 2 weeks + keep logs; Verbal feedback HF nurse
  Arms: Condition 8

SUMMARY:
The aim of this study is optimize the STAR (SympTom mAnagement self-caRe) intervention to support patients with HF in staying healthy, and particularly in self-monitoring and managing symptoms. The STAR intervention includes promising components aiming at improving patient outcomes in terms of interference of bothersome symptoms, self-care, quality of life (QoL) and healthcare utilization.

In this study, the intervention components are tested in an optimization trial in 320 patients with HF from 8 HF clinics in the Netherlands. This study will result in an optimized STAR intervention, composed of the best components, that is effective, scalable, and efficient to improve patient outcomes and can be used in HF clinics.

DETAILED DESCRIPTION:
According to the Multiphase Optimization StraTegy (MOST), in this optimization trial, the investigators aim to evaluate and optimize the components of the STAR intervention prior to evaluation in an RCT. The STAR intervention consists of different components (modules): one basic module and three key modules. The basic module consists of information about HF and preparatory exercises; the key modules consist of training to improve symptom awareness, symptom management counseling, and symptom management option experiments. Following MOST, the investigators developed different intensity version of each key module: a low intensity version and a high intensity version. The low intensity version is more basic compared to the high intensity version. The low and high intensity versions differ in the mode of feedback from the HF nurses (written vs verbal) or intensity of exercises or feedback (e.g. one week vs two weeks); the content remains the same. These two versions allow the investigators to evaluate which mode and dose works best for each module and are tested in this optimization trial using factorial experiments. The most contributing versions of modules are then integrated into the STAR intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HF (irrespective of ejection fraction) and symptomatic NYHA class II or III.
* 18 years or older.
* Willing and able to provide written informed consent.
* Life expectancy >6 months.
* Optimal medical HF treatment following ESC HF guidelines (i.e. 'patients with stable HF').

Exclusion Criteria:

* Participants living in a care facility (e.g. nursing home, revalidation center).
* Language barrier preventing sufficient understanding and communication in Dutch.
* Participants who are hospitalized during inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Interference of bothersome symptoms | From Baseline (T0) to the end of the last module (T4) at the following time points: Baseline (T0), week 1 (T1), week 2-3 (T2), week 4 (T3), week 6 (T4)
  For interference of bothersome symptoms three domains of the Kansas City Cardiomyopathy Questionnaire will be assessed: symptom, physical function and symptom stability.
  Scores are standardized on a scale from 0 to 100, with higher scores representing fewer symptoms.

SECONDARY OUTCOMES:
Self-care | Measured at baseline and week 6 (T4)
  Using the Self-Care Heart Failure Index version 7.2, scales self-care maintenance, symptom perception, and self-care management. Scores range from 0-100, scores higher than 70 indicate better self-care.
HRQoL | Measured at baseline and week 6 (T4)
  The 23-item Kansas City Cardiomyopathy Questionnaire will be used to evaluate the Health related Quality of life of patients with HF. The items are divided into five domains: physical limitations, social limitations, symptoms, self-efficacy, and quality of life.
  Scores are standardized on a scale from 0 to 100, higher scores represent fewer symptoms and better overall health status.
Healthcare utilization | Measured at baseline and week 6 (T4)
  Using hospital data: number of HF-related ER and hospital admissions
Healthcare utilization 2 | Measured at baseline and week 6 (T4)
  Using hospital data: Length of stay in days
Healthcare utilization 3 | Measured at baseline and week 6 (T4)
  Using hospital data: Number of unscheduled (telephone) consultations with the HF outpatient clinic).

OTHER OUTCOMES:
Illness perceptions | Measured at week 1 (T1) and week 2-3 (T2 )
  Illness perception will be measured with the 8-item Brief-Illness perception Questionnaire, assessing patients' cognitive and emotional representations of illness. The score range is 0-80. Higher scores indicate worse illness perception.
HF knowledge | Measured at baseline and week 1 (T1)
  15-item Dutch Heart Failure Knowledge Scale will be used to measure HF knowledge in general, HF treatment, and HF symptoms and symptom recognition. Range of score is 0-15, with higher scores representing optimal knowledge.
Interoception | Measured at baseline, week 1(T1), week 2-3 (T2), week 6 (T4)
  The 37-item Multidimensional Assessment of Interoceptive Awareness version 2 will be used to measure eight dimensions of interoception (noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, trust). Scale scores are 0-5, where higher scores indicate more interoceptive awareness.
Symptom attribution | week 2-3 (T2)
  The Illness Perception Questionnaire (revised) identity scale will be used to measure symptom attribution. Participants will be asked if they have experienced a number of symptoms since their illness, and if they feel the symptoms are related to their current illness. Response is by answering 'yes' or 'no' to each symptom. The number of yes-rated items are summed to give an overall score (range 0- 21). A high score represents strongly held beliefs about the number of symptoms attributed to HF.
Confidence, and symptom management skills | Measured at week 2-3 (T2) and at week 6 (T4)
  Confidence will be measured using the 10-item Self Care Self-Efficacy Scale measuring self-care self-efficacy in chronic illness. The standardized score range from 0-100. Scores >70 indicate better self-care confidence.
Symptom management skills | Measured at week 4 (T3) and week 6 (T4)
  Symptom management skills will be evaluated with 8-item Control Attitudes Scale-Revised. Range score is 8-40, higher scores indicate greater perceived control.
User logs (patients and nurses) | Measured at week 1 (T1), week 2-3 (T2), week 4 (T3), week 6 (T4)
  Treatment fidelity will be evaluated with the user logs of the platform of patient and nurse. Written feedback from HF nurses to patients in each module will be evaluated using self-assessments for the HF nurses. The number of minutes of the verbal feedback in each module will be registered by nurses.
Self-assessments | Measured at week 4 (T3)
  Descriptive analysis of self-assessments made by patients in module 2.
User experiences | Measured at the end of the intervention week 7-8
  Experiences of patients will be evaluated using semi-structured interviews. We aim to include 5 participants per version per module (total 40 participants). All participating HF nurses are asked to share their experiences with the research team at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Heleen Westland, PhD, Principal Investigator — UMC Utrecht; Tiny Jaarsma, PhD, Study Chair — UMC Utrecht and Linköping University

IPD SHARING:
Plan to Share IPD: No
Interested parties can request access to this data-set via our institutional data access committee (DC) for the EGA; based on the assessment of the DAC access to this data-set will be granted or declined.